CLINICAL TRIAL: NCT03528005
Title: Effectiveness of Integrated Care Network for Community-living Older Adults: a Randomized-Controlled Trial
Brief Title: Effectiveness of Integrated Care Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Liang-Kung Chen, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM107042F
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Fragility; Multimorbidity
Keywords: Integrated Health Care Systems; Multimorbid; Multi-domain intervention; Clinical Trials, Randomized

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): A regular health education program was provided by case managers only.
- Intervention (Experimental): Multi-domain intervention included exercise,cognitive training, diet education, and disease consultation was conducted for two hours twice per week in the first month, once per week in the second month, and once per month since third month.
  Interventions: Behavioral: Multi-domain intervention

INTERVENTIONS:
Behavioral: Multi-domain intervention — 60 minutes cognitive training, 45 minutes physical exercise, 15 diet nutrition and intermittent disease management consultation
  Arms: Intervention

SUMMARY:
This project aims to examine the effectiveness of the community-based integrated care service model , based on a multi-domain intervention program, among community-dwelling older adults. Moreover, the investigators use the value-based healthcare standard set as well as comprehensive geriatric assessment as outcome measures and to use the randomized controlled trial design to validate the clinical effectiveness.

DETAILED DESCRIPTION:
Population aging and the progress of medical technology are two main causes for the increase of healthcare expenditure. Effective management of medical expenditure and maintenance of health care quality have become the most important task for the public health and clinical care services. Both United Kingdom and the World Health Organization proposed introducing interdisciplinary team care to improve health of older people and to maximize their independence. Prof Michael Porter has addressed the current difficulty of healthcare system, and proposed that healthcare system should pursuit long-term outcome to promote the value of health care. This project aims to echo the international trends, using Taiwan healthcare system as the basis to establish the community-based integrated care service model, and to use the randomized controlled trial design to validate the clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* age ≧ 65 years
* three or more chronic conditions, defined by National Health Insurance list of chronic conditions
* covered by National Health Insurance

Exclusion Criteria:

* could not understanding protocol or communication with research nurses
* malignant diseases under active treatments
* life expectancy less than twelve months
* admitted in the long term facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 398 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Changes from baseline life quality at 3, 6, 9, 12 month | baseline, 3, 6, 9, 12 month
  measured by the 36-Item Short Form Health Survey (SF-36).

SECONDARY OUTCOMES:
Changes from baseline standard set of health outcome measures for older persons at 3, 6, 9, 12 month | baseline, 3, 6, 9, 12 month
  a standard health care set proposed by the International Consortium for Health Outcomes Measurement (ICHOM)

OTHER OUTCOMES:
Changes from baseline high sensitive C-Reactive Protein in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline high sensitive C-Reactive Protein in mg/dl at sixth and twelfth month
Changes from baseline total cholesterol in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline total cholesterol in mg/dl at sixth and twelfth month
Changes from baseline triglycerides in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline triglycerides in mg/dl at sixth and twelfth month
Changes from baseline HDL-C in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline High-density lipoproteins (HDL) in mg/dl at sixth and twelfth month
Changes from baseline LDL-C in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline Low-density lipoproteins (LDL) in mg/dl at sixth and twelfth month
Changes from baseline fasting glucose in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline fasting glucose in mg/dl at sixth and twelfth month
Changes from baseline HbA1c in % at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline Hemoglobin A1c in % at sixth and twelfth month
Changes from baseline insulin in mIU/L at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline insulin in mIU/L at sixth and twelfth month
Changes from baseline uric acid in mg/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline uric acid in mg/dl at sixth and twelfth month
Changes from baseline body mass index in kg/m^2 at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline body mass index in kg/m^2 at sixth and twelfth month
Changes from baseline albumin in g/dl at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline albumin in g/dl at sixth and twelfth month
Changes from baseline Vitamin D in ng/ml at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline Vitamin D in ng/ml at sixth and twelfth month
Changes from baseline Vitamin B12 in pg/ml at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline Vitamin B12 in pg/ml at sixth and twelfth month
Changes from baseline homocysteine in micromol/l at sixth and twelfth month | baseline, 6,12 month
  Changes from baseline homocysteine in micromol/l at sixth and twelfth month

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD.PhD., Study Director — Aging and Health Research Center, National Yang Ming University
Locations (6):
- Taiwan (6):
  - Hualien Tzu Chi Hospital,Buddhist Tzu Chi Medical Foundation, Hualien City
  - Shulin Primary Care center, New Taipei City
  - Yingge Primary Health Care center, New Taipei City
  - Cheng's primary care clinic, New Taipei City
  - National Yang-Ming University Hospital, Yilan
  - Taipei Veterans General Hospital Yuanshan Branch, Yilan

REFERENCES:
- [Derived] Lee WJ, Peng LN, Lin MH, Kim S, Hsiao FY, Chen LK. Enhancing Intrinsic Capacity and Related Biomarkers in Community-Dwelling Multimorbid Older Adults Through Integrated Multidomain Interventions: Ancillary Findings From the Taiwan Integrated Geriatric (TIGER) Trial. J Am Med Dir Assoc. 2024 May;25(5):757-763.e4. doi: 10.1016/j.jamda.2023.10.006. Epub 2023 Nov 7. PMID 37949432
- [Derived] Lee WJ, Peng LN, Lin CH, Chen RC, Lin SZ, Loh CH, Kao SL, Hung TS, Chang CY, Huang CF, Tang TC, Huang ST, Wen YW, Hsiao FY, Chen LK; Taiwan Integrated Geriatric Care Study Group. Effects of incorporating multidomain interventions into integrated primary care on quality of life: a randomised controlled trial. Lancet Healthy Longev. 2021 Nov;2(11):e712-e723. doi: 10.1016/S2666-7568(21)00248-8. Epub 2021 Oct 22. PMID 36098028